CLINICAL TRIAL: NCT01354119
Title: Long-term Benefit of Aortic Stent-graft in Patients With Distal Aortic Dissection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough participants enrolled
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Min Song, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADdistal_graft
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Aortic Dissection; Aortic Aneurysm; Stent-graft
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early intervention (Active Comparator): Early intervention: stent-graft just after acute phase
  Interventions: Procedure: Aortic stent-graft
- Conservative (No Intervention): Conservative: medial follow-up without early intervention

INTERVENTIONS:
Procedure: Aortic stent-graft — Early intervention with aortic stent-graft
  Arms: Early intervention

SUMMARY:
Background: Aortic stent-graft is useful to occlude intimal tear and prevent further dilatation of the false lumen in patients with aortic dissection. The long-term benefit of aortic stent-graft in patients with uncomplicated distal aortic dissection has not been well demonstrated, especially in patients at high risk of aneurysmal change and death.

Purpose: The purpose of the study is to evaluate long-term clinical benefit of stent-graft insertion performed just after the acute phase into the descending thoracic aorta in patients with distal aortic dissection and at high risk of aneurysmal change of the dissected aorta.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated distal aortic dissection
* Initial false lumen diameter >= 22 mm

Exclusion Criteria:

* Old age (> 75 years old)
* Other comorbidity or malignancy with life expectancy < 5 years
* Complicated dissection requiring aortic surgery or intervention
* Sudden death in acute phase
* Marfan syndrome

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Aortic aneurysm and death | 4 years

SECONDARY OUTCOMES:
Events and complications | 4 years
  paraplegia cerebrovascular accident aorta surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea